CLINICAL TRIAL: NCT00217347
Title: Evaluation of Efficiency of Esophageal Capsule Endoscopy in the Screening of Patients With Gastroesophageal Reflux Disease or Dyspepsia as Compared to Upper Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD/05/3-J
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Gastroesophageal Reflux Disease; Dyspepsia
Keywords: Gastroesophageal reflux; Dyspepsia; Esophageal Capsule Endoscopy
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia | interventions — Endoscopy

INTERVENTIONS:
Device: Esophageal Capsule Endoscopy

SUMMARY:
The exploration of evocative symptoms of esophageal reflux disease or dyspepsia is based on a relatively invasive endoscopic examination, often badly tolerated, and which, in France, is carried out in 50% of the cases under general anaesthesia. The development of a Capsule Endoscopy, of single use, of esophageal exploration (PILLCAM OESO), could allow a painless exploration of the oesophagus, without infectious risk.The aim of this study is to validate the information provided by the Esophageal Capsule Endoscopy compared to upper endoscopy in the screening of patients with gastroesophageal reflux disease or dyspepsia . For that these patients, after being informed and to have given their signed assent, will initially have an exploration by Esophageal Capsule Endoscopy and then, the very same day or within 3 days maximum, a upper endoscopy'. The information provided by the Esophageal Capsule Endoscopy then by the upper endoscopy will be analyzed by investigators different. This study should make it possible to evaluate the parameters of specificity, sensitivity and predictive values of Esophageal Capsule Endoscopy in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Patient age is 18 years or older
* Patient Suffers from gastroesophageal reflux disease or dyspepsia, did not undergo previous upper endoscopy, with clinical indication to upper endoscopy,able to tolerate an upper endoscopy without general anesthesia
* Patient agrees and signs the Informed Consent Form

Exclusion Criteria:

* Dysphagia
* Known Zenker's Diverticulum
* Known or suspected intestinal obstruction.
* Cardiac pacemakers or other implanted electro medical devices.
* Female pregnant patient
* Upper Endoscopy for control or recent upper endoscopy
* Chronic alcoholism defined by a daily consumption of alcohol over 80 g
* Severe hepatopathy
* Severe, primitive or secondary gastroparesis
* Known cancer
* Abnormalities of coagulation
* Incapacity to understand and sign a sensible consent of participation to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To determine the parameters of sensitivity, specificity, positive and negative predictive values of the Esophageal Capsule Endoscopy

SECONDARY OUTCOMES:
To compare Esophageal Capsule Endoscopy and upper endoscopy in detection and classification of esophagitis.
To determine the inter-observer agreement for the classification of esophagitis.
To compare Esophageal Capsule Endoscopy and upper endoscopy in detection of stomachal or duodenal lesions.
To evaluate the tolerance of the two examinations

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul Galmiche, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France